CLINICAL TRIAL: NCT06091904
Title: Effects of Sufentanil on the Intraoperative Hemodynamic Parameters in Patients Undergoing Extracranial-intracranial Bypass Surgery: a Prospective Randomized Controlled Trial
Brief Title: Effects of Sufentanil on the Intraoperative Hemodynamics
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Chang-Hoon Koo, Assistant professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Bypass-SFTN
Record Dates: First submitted 2023-10-13; First posted 2023-10-19 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Intraoperative Hypotension
MeSH Terms: interventions — Sufentanil; Remifentanil

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- sufentanil group (Experimental): sufentanil is administered for analgesic during general anesthesia
  Interventions: Drug: Sufentanil
- remifentanil group (Active Comparator): remifentanil is administered for analgesic during general anesthesia
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Sufentanil — Induction: sufentanil TCI 0.3 ng/ml Maintenance: sufentanil TCI 0.05-0.5 ng/ml
  Arms: sufentanil group
Drug: Remifentanil — Induction: remifentanil TCI 3 ng/ml Maintenance: remifentanil TCI 0.5-5 ng/ml
  Arms: remifentanil group

SUMMARY:
This study is a randomized, controlled trial. A total of 92 patients will be randomized to receive sufentanil or remifentanil during extracranial-intracranial bypass surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergo elective extracranial-intracranial bypass surgery
* American Society of Anesthesiologists grade 1,2,3
* Age > 18 years old

Exclusion Criteria:

* Refuse to participate to the study
* American Society of Anesthesiologists grade 4
* Body Mass Index < 18.5 kg/m2 or > 35 kg/m2
* Allergic history of opioid
* pregnant
* MAO Inhibitor user
* Severe respiratory insufficiency

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2023-11-24 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Intraoperative hypotension | During surgery
  MAP < 80 mmHg

SECONDARY OUTCOMES:
Inotropic requirements | During surgery
  cumulative doses of inotropics during surgery
Incidence of bradycardia | During surgery
  heart rate < 40/min
Incidence of tachycardia | During surgery
  heart rate > 100/min
Maximum systolic blood pressure | During surgery
  maximal systolic blood pressure
Minimum systolic blood pressure | During surgery
  minimal systolic blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Hoon Koo, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No